CLINICAL TRIAL: NCT03607942
Title: Use of a Liquid Supplement Containing 2 Human Milk Oligosaccharides (HMOs) in Preterm Infants: a Double-blind, Randomized, Controlled Trial
Brief Title: Use of a Liquid Supplement Containing 2 Human Milk Oligosaccharides (HMOs) in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17.02.INF
Record Dates: First submitted 2018-04-05; First posted 2018-07-31 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Formula (Experimental): The experimental group will receive a liquid supplement containing 2 specific HMOs
  Interventions: Dietary Supplement: HMO supplement
- Control Formula (Placebo Comparator): The control group will receive a liquid placebo
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: HMO supplement — HMO supplement will be given three times a day, not mixed with any feeding.
  Arms: Experimental Formula
Dietary Supplement: Placebo comparator — Control product without any HMOs. The Placebo Comparator will be matched to the experimental product in energy content.
  Arms: Control Formula

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled trial in preterm infants conducted at least 4 centers in France, consisting of 2 parallel groups. The experimental group will receive a neonatal supplement containing 2 specific HMOs. The control group will receive a placebo neonatal supplement that does not contain any HMOs, but matched to the experimental product in energy content.

This study will include a total of approximately 86 male and female preterm infants born between 27 and 32 weeks' gestational age with birth weight ≤1700 g, who are younger than 7 days of age.

The primary objective of the study is to demonstrate the safety and tolerance of HMOs in preterm infants by monitoring weight gain rates in both of the two randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* Infant's birth weight ≤1700 g.
* Infant's gestational age ≥ 27 weeks + 0 days and ≤ 32 weeks + 6 days.
* Infant is clinically stable
* Infants are eligible to start HMOs / placebo as soon as possible after birth, but still within the first 7 days of life.
* Written informed consent has been obtained from the parents/legally acceptable representative (LAR).

Exclusion Criteria:

* Parents not willing / not able to comply with the requirements of study protocol.
* Infants receiving ongoing prophylactic antifungal therapies.
* Infants experiencing early onset sepsis.
* Major congenital or chromosomal abnormality known to affect growth.
* Liver failure.
* Severe intrauterine growth restriction (IUGR) as defined by having birth weight less than 2nd percentile on the Fenton growth chart.
* Peri-/intra-ventricular haemorrhage (grade 3-4 in Papille classification) .
* Infant in critical condition needing intubation or inotropic agents for treatment.
* Infant requiring prolonged (more than 3 doses) of steroid treatment.
* Infants' participation in another interventional clinical trial that would have significant impact on current study's results.
* Infants who have already achieved Full Enteral Feeding (FEF) prior to enrolment, using the definition accepted by neonatal unit as per standard practice (150 mL/kg/day).

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Feeding tolerance | Change from Full Enteral Feeding (FEF) Day 1 (start of FEF defined as achieving 150ml/day/kg of enteral feeding and discontinuation of parenteral feeding) and FEF Day 21 (approximately 5 weeks after enrollment)
  The primary objective is to demonstrate non-inferiority in feeding tolerance (defined as number of days to reach full enteral feeding) of preterm infants receiving a liquid supplement composed of 2 HMOs compared to those receiving the placebo.

SECONDARY OUTCOMES:
Length | Change from enrolment (baseline) (if feasible) through study completion, average of 4 months
  Through standardized measurement for neonates
Head circumference | Change from enrolment (baseline) (if feasible) through study completion, average of 4 months
  Through standardized measurement for neonates
Weight gain | Change from enrolment (baseline) (if feasible) through study completion, average of 4 months
  Through standardized measurement for neonates
Assessment of infant illnesses and infections | Change from enrolment (baseline) (if feasible) through study completion, average of 4 months
  Through Adverse Event reporting
Tolerance to feeding regimen | Change from enrolment (baseline) (if feasible) through study completion, average of 4 months
  Through neonatal unit records
Physical signs of gastrointestinal tolerance | Change from enrolment (baseline) (if feasible) through study completion, average of 4 months
  Through neonatal unit records
Breast milk composition such as energy, carbohydrate, proteins and fats using mid-infrared transmission methods | Change from enrolment (baseline) (if feasible) until FEF Day 21, average of 5 weeks
  Macro and micro nutrients
Standard Adverse Event reporting for safety assessment | Change from enrolment (baseline) (if feasible) through study completion, average of 4 months
  Through investigator-confirmed Adverse Event reporting
Fecal microbiota composition and diversity | Change from enrolment (baseline) through two-months corrected age visit
  Fecal microbiota composition and diversity will be assessed using next generation shotgun metagenomics sequencing to provide taxonomic composition and diversity metrics. Quantifiable changes from baseline and between feeding groups in absolute concentrations of bifidobacteria will be assessed using quantifiable polymerase chain reaction
Fecal metabolic profile | Change from enrolment (baseline) through two-months corrected age visit
  Measures of fecal metabolism will include fecal power of hydrogen (pH) and fecal organic acids (including lactate, propionate, butyrate, acetate, isobutyrate, isovalerate, valerate, formic acid, hexanoic acid, caprylic acid, capric acid, pelargonic acid, undecanoic acid, dodecanoic acid and total fecal organic acids).
Markers for gut health, gut maturation and immune status | Change from enrolment (baseline) (if feasible) until FEF Day 21
  Markers for gut health, gut maturation and immune status will be assessed through measures of:
  Fecal level of calprotectin, alpha 1 antitrypsin, pancreatic elastase, human beta-defensin 2 , secretory immunoglobulin A, Plasma level of citrulline and twenty four additional Amino Acids Urinary levels of intestinal fatty acid binding protein
Early life development outcomes | At 12 Months Corrected age Visit, 18 Months Corrected age Visit, and 24 Months Corrected age Visit
  Aligned with standard routine care, post-discharge clinical assessments of preterm infants include clinically relevant events since last visit, feeding practice (complementary feeding, adequate food intake), Gastrointestinal-related symptoms (sleep, crying), somatic examination (physical examination of skin, digestion, abdomen, hip), Neurosensory Examination (hearing / visual function, gross motor), Relationship and Communication Development (normal or abnormal communication, neurological or psychomotor examination, relationship
  / behavior disorders). All clinical assessments will be standardized across sites. Ages and Stages Questionnaire-3 will be administered to parents to assess their report of child's developmental progress based on Communication, Gross Motor, Fine Motor, Problem Solving, and Personal-Social domains.
Cognitive development outcomes | 24 Months Corrected age Visit
  Will be assessed through the composite scores or scale scores of the Bayley Scales of Infant and Toddler Development - Third Edition (Bayley-III)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Hascoët, Prof, Study Director — CHRU Nancy
Locations (7):
- France (7):
  - CHU de Bordeaux - Hôpital des Enfants, Bordeaux
  - Hôpital Couple Enfant, Grenoble
  - Hôpital Nord, Marseille
  - Maternité Régionale Universitaire A. Pinard - CHRU Nancy, Nancy
  - Hôpital femme-maternité, Nantes
  - CHR Orléans - Hôpital de la Source, Orléans
  - Centre Hospitalier de Pau, Pau

IPD SHARING:
Plan to Share IPD: No